CLINICAL TRIAL: NCT00560911
Title: Impact of Self-Management of Oral Anticoagulation in the Elderly in Terms of Mortality and Morbidity: a Randomized Controlled Trial - SPOG 60+
Brief Title: Major Outcomes in Elderly Patients With Self-Management of Oral Anticoagulation (SPOG60+)
Acronym: SPOG60+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Boehringer Mannheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SPOG60+
Record Dates: First submitted 2007-11-17; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Long-Term Oral Anticoagulated Patients
Keywords: oral anticoagulation; self-management; elderly patients; randomised controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1Self-management (Other)
  Interventions: Behavioral: educational program for the self-management of OAC
- 2 Routine control (Other)
  Interventions: Behavioral: 1 hour education - afterwards physician leaded OAC control

INTERVENTIONS:
Behavioral: educational program for the self-management of OAC — Patients in the self-management group participated in 4 consecutive weekly instruction sessions of 90 to 120 minutes each, in groups of 3 to 6 patients.
  After participation in the structured programme, the patients were encouraged to control their INR values by self-monitoring once a week and to adjust their anticoagulant dosage accordingly.
  Arms: 1Self-management
Behavioral: 1 hour education - afterwards physician leaded OAC control — Patients in the routine control group participated a single 90-minute session
  During the whole study period, they were advised with regard to changes in the anticoagulant dosage by their usual attending physicians, either in general practice or at a hospital-based specialised anticoagulation clinic.
  Arms: 2 Routine control

SUMMARY:
Self-management is safe and reliable in patients with long-term oral anticoagulation (OAC). However, no study has yet assessed the safety and efficacy of OAC self-management in elderly patients with major thromboembolic and haemorrhagic complications as primary outcomes.

In this multi-centre, open, randomised controlled trial, patients aged 60 years or will be randomised into a self-management or routine care group and followed up for at least two years.

The primary hypothesis of the study is that self-management of oral anticoagulation is superior compared to routine control in terms of reducing thromboembolic events requiring hospitalisation and all major bleeding complications as the primary endpoint.

DETAILED DESCRIPTION:
Oral anticoagulation (OAC) has been shown to be highly effective in preventing thromboembolic complications in patients for whom it is indicated. Numerous studies have documented that elderly patients seem to benefit most from OAC therapy. Atrial fibrillation (AF), the incidence of which increases with age and approaches 10% for individuals aged ≥ 80 years, carries the main risk for stroke, and among elderly patients without antithrombotic therapy,

Despite its proven benefit, numerous studies have reported reluctance in prescribing OAC due to a variety of barriers, especially in the elderly. Risk of haemorrhage, which is in fact twice as great in those over 70 years of age as in younger patients, is one of the major determinants of refusal to prescribe OAC therapy. The risk of stroke rises steeply in patients with atrial fibrillation when INR values are less than 1.8 and INR values greater than 4 to 5 are rapidly associated with increased bleeding rates. Due to relatively small therapeutic ranges, the reality is often that only a small percentage of the INR values have been found to be within the target range, which can be low as 29% of INR measurements, as seen in routine care patients prior to participation in a randomised self-management programme study.

One way to improve OAC care is by introducing patients' self-management of OAC therapy. In this context it is important to differentiate between INR self-testing alone, and full self-management. Self-management includes self-adaptation of the anticoagulation treatment based on self-monitoring results after the patients have participated in a structured instruction and treatment programme.

Our study aims to provide answers to this important medical question by examining elderly patients receiving long-term anticoagulation treatment and randomised into self-management versus routine-care groups, with thromboembolic and haemorrhagic complications as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* long-term anticoagulation
* either with phenprocoumon or acenocoumarol
* age ≥ 60 years
* written informed consent

Exclusion Criteria:

* previous participation in a self-management OAC programme
* severe cognitive
* terminal illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2002-03; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
combined endpoint of all thromboembolic events requiring hospitalisation and all major bleeding complications | during the time of follow up (at least two years)

SECONDARY OUTCOMES:
frequency and duration of hospitalisation | during the time of follow up (at least two years)
mortality | during the time of follow up (at least two years)
recurrence of stroke | during the time of follow up (at least two years)
numbers of INR values above 4.5 or lower than 1.7 | during the time of follow up (at least two years)
treatment-related quality of life analysis | during the time of follow up (at least two years)
cost-effectiveness evaluations | during the time of follow up (at least two years)
median of squared INR value deviation (INR - ½(Upper Value of Target INR Range + Lower Value of Target INR Range)) | during the time of follow up (at least two years)
percentage of individual patients' INR values within the target range and the percentage of time within target range | during the time of follow up (at least two years)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Didjurgeit, psychologist, Principal Investigator — DIeM - Institute for Evidence-based Medicine, Cologne, Germany; Andrea Siebenhofer, consultant, Study Chair — Department of Internal Medicine, Medical University of Graz, Austria
Locations (3):
- Austria (2):
  - Medical University Graz, Graz, Styria
  - Medical University of Vienna, Vienna
- DIeM - Institute for Evidence-based Medicine, Cologne, Germany

REFERENCES:
- [Result] Siebenhofer A, Rakovac I, Kleespies C, Piso B, Didjurgeit U. Self-management of oral anticoagulation in the elderly: rationale, design, baselines and oral anticoagulation control after one year of follow-up. A randomized controlled trial. Thromb Haemost. 2007 Mar;97(3):408-16. PMID 17334508